CLINICAL TRIAL: NCT04276831
Title: Comparison of Cardiovascular Response and Ease of Intubation Using Laryngoscope McCoy With Macintosh in Malay Race in Indonesia
Brief Title: Comparison Between Laryngoscope McCoy With Macintosh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Riyadh Firdaus, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IndonesiaUAnes046
Record Dates: First submitted 2020-01-08; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Surgery
Keywords: Intubation; Cardiovascular response; Laryngoscope

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngoscope McCoy (Active Comparator): Patients will be intubated using laryngoscope McCoy
  Interventions: Device: Laryngoscope McCoy
- Laryngoscope Macintosh (Active Comparator): Patients will be intubated using laryngoscope Macintosh
  Interventions: Device: Laryngoscope Macintosh

INTERVENTIONS:
Device: Laryngoscope McCoy — Subjects who fulfill inclusion criteria will be intubated using laryngoscope McCoy
  Arms: Laryngoscope McCoy
Device: Laryngoscope Macintosh — Subjects who fulfill inclusion criteria will be intubated using laryngoscope Macintosh
  Arms: Laryngoscope Macintosh

SUMMARY:
This study aimed to compare cardiovascular response and ease of intubation using laryngoscope McCoy with Macintosh

DETAILED DESCRIPTION:
Eighty-two subjects were given informed consent before enrolling the study and randomized into two groups: McCoy and Macintosh. Non-invasive blood pressure

ELIGIBILITY:
Inclusion Criteria :

* adults (18 - 65 years old)
* body mass index 18,5 - 30 kg/m2
* physical status with ASA 1 -2
* patients who agreed to participate in this study and sign informed consent.

Exclusion Criteria:

* pregnancy
* history of infarct miocard
* right or left heart failure
* P-R interval 0,24 seconds
* heart block degree 2 or 3
* using pace maker
* history of cerebrovascular disease
* tachycardia or bradycardia
* on medication (antiarrhythmic drugs, beta blocker, heart stimulant)
* suspect difficult airways
* including ventilation (assesment with MOANS) or intubation (assesment with LEMONS)
* patients with increase of intracranial pressure (e.g.head injury)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Measurement of systolic blood pressure | 3 minutes
  Measurement of systolic blood pressure by using automated sphygmomanometer and recorded in mmHg
Measurement of diastolic blood pressure | 3 minutes
  Measurement of diastolic blood pressure by using automated sphygmomanometer and recorded in mmHg
Measurement of mean arterial pressure | 3 minutes
  Measurement of mean arterial pressure by using automated sphygmomanometer and recorded in mmHg
Measurement of heart rate | 3 minutes
  Measurement of heart rate and recorded beats per minute

SECONDARY OUTCOMES:
Concentration of opioid administration for 24 hours after surgery | 24 hours
  Concentration of opioid administration in mcg

CONTACTS AND LOCATIONS:
Overall Officials: Riyadh Firdaus, MD, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xue FS, Wang Q, Liao X, Yuan YJ. Cardiovascular intubation responses with Airway Scope and Macintosh laryngoscope. Anaesthesia. 2012 Apr;67(4):434-5; author reply 435-6. doi: 10.1111/j.1365-2044.2012.07071_1.x. No abstract available. PMID 22409804
- [Result] Randell T. Haemodynamic responses to intubation: what more do we have to know? Acta Anaesthesiol Scand. 2004 Apr;48(4):393-5. doi: 10.1111/j.1399-6576.2004.00381.x. No abstract available. PMID 15025596
- [Result] Shimoda O, Ikuta Y, Isayama S, Sakamoto M, Terasaki H. Skin vasomotor reflex induced by laryngoscopy: comparison of the McCoy and Macintosh blades. Br J Anaesth. 1997 Dec;79(6):714-8. doi: 10.1093/bja/79.6.714. PMID 9496201
- [Result] Bilgin H, Bozkurt M. Tracheal intubation using the ILMA, C-Trach or McCoy laryngoscope in patients with simulated cervical spine injury. Anaesthesia. 2006 Jul;61(7):685-91. doi: 10.1111/j.1365-2044.2006.04706.x. PMID 16792615
- [Result] Noppens RR, Geimer S, Eisel N, David M, Piepho T. Endotracheal intubation using the C-MAC(R) video laryngoscope or the Macintosh laryngoscope: a prospective, comparative study in the ICU. Crit Care. 2012 Jun 13;16(3):R103. doi: 10.1186/cc11384. PMID 22695007